CLINICAL TRIAL: NCT05384951
Title: β-hydroxy-β-methylbutyrate (HMB) Pilot Feasibility and Efficacy Study in Cerebral Palsy (CP)
Brief Title: HMB Cerebral Palsy Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gillette Children's Specialty Healthcare (Other)
Collaborators: University of Minnesota (Other); Metabolic Technologies, LLC (Unknown)
Responsible Party: Principal Investigator, Elizabeth Boyer, Clinical Scientist, Gillette Children's Specialty Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00015262
Record Dates: First submitted 2022-05-02; First posted 2022-05-23 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy
Keywords: HMB; Vitamin D; Safety; Compliance; Strength; Muscle Mass; Mobility; β-hydroxy-β-methylbutyrate; Calcium β-hydroxy-β-methylbutyrate
MeSH Terms: conditions — Cerebral Palsy; Patient Compliance | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Single group repeated measures design with 12 weeks of no intervention (control period) followed by 12 weeks of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HMB + Vitamin D3 Supplement (Experimental): Supplement delivery will be a tablet containing both HMB & Vitamin D3. HMB will be administered in its calcium salt form. One tablet will contain 750 mg HMB + 250 IU of Vitamin D3. The target dosage is 3 g HMB + 1000 IU of Vitamin D3 per day.
  Interventions: Dietary Supplement: HMB + Vitamin D3

INTERVENTIONS:
Dietary Supplement: HMB + Vitamin D3 — The supplement will be taken orally twice daily. Participants will take 2 blended HMB + Vitamin D3 tablets in the morning and 2 tablets in the evening for 12 weeks.

SUMMARY:
This is a pilot study of β-hydroxy-β-methylbutyrate (HMB) + Vitamin D3 supplementation in adolescents with cerebral palsy. The primary objective is to quantify safety, compliance, and acceptability of daily combined HMB + Vitamin D3 supplementation for 12 weeks in adolescents with CP. The secondary objective is to quantify changes in lower extremity muscle mass, strength, and functional mobility after daily combined HMB + Vitamin D3 supplementation for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cerebral palsy
* Spastic or mixed tone
* GMFCS Level I-III (i.e., ambulatory)
* 13-17 years old
* Physical training level expected to remain relatively constant over the study period
* Ability to follow directions, including swallowing multiple pills daily and complying with reproductive risk recommendations (post-menarchal females)
* Within reasonable driving distance to the University of Minnesota - Twin Cities
* Reads English

Exclusion Criteria:

* Pregnant, lactating, or trying to become pregnant
* Surgery in the past 9 months
* Botulinum toxin injections in past 3 months
* Selective dorsal rhizotomy in the past 12 months
* Upcoming invasive treatment within the study period that may affect strength or functional mobility (e.g., surgery, botulinum toxin injections, intrathecal baclofen pump or dosage change)
* Liver disease or liver disorder
* Kidney disease or disorder
* Prescription drug or nutrition supplement contraindications
* Excessive research or medical-related radiation exposure in the past 12 months (approximately 500 mrem or greater)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the incidence of Treatment-Emergent Adverse Events with supplementation as assessed by renal (kidney) function - specific gravity | Pre-supplementation (12 wks), post-supplementation (12 wks)
  Specific gravity will be measured via urinalysis with microscopy (unitless; ratio of urine density [g/cm^3] divided by density of pure water).
Difference in the incidence of Treatment-Emergent Adverse Events with supplementation as assessed by renal (kidney) function - pH | Pre-supplementation (12 wks), post-supplementation (12 wks)
  pH will be measured via urinalysis with microscopy (usually presented unitless; moles H+ per liter).
Difference in the incidence of Treatment-Emergent Adverse Events with supplementation as assessed by renal (kidney) function - microscopy | Pre-supplementation (12 wks), post-supplementation (12 wks)
  Molecular concentrations in urine will be measured via urinalysis with microscopy. The following molecular concentrations will be measured: total protein, glucose, ketones, blood, bilirubin, and urobilinogen (all units: unitless).
Difference in the incidence of Treatment-Emergent Adverse Events with supplementation as assessed by renal (kidney) function - BUN | Pre-supplementation (12 wks), post-supplementation (12 wks)
  Blood urea nitrogen (BUN; units: mg/dL) will be measured using a blood sample.
Difference in the incidence of Treatment-Emergent Adverse Events with supplementation as assessed by renal (kidney) function - creatinine | Pre-supplementation (12 wks), post-supplementation (12 wks)
  Creatinine will be measured using a blood sample. It will be used to estimate glomerular filtration rate (mL/min/m^2 body surface area).
Difference in the incidence of Treatment-Emergent Adverse Events with supplementation as assessed by hepatic (liver) function - enzymes | Pre-supplementation (12 wks), post-supplementation (12 wks)
  Hepatic enzyme function will be measured with a blood sample. Outcomes include alkaline phosphatase [ALP], aspartate aminotransferase [AST], alanine aminotransferase [ALT] (all units: units per liter).
Difference in the incidence of Treatment-Emergent Adverse Events with supplementation as assessed by hepatic (liver) function | Pre-supplementation (12 wks), post-supplementation (12 wks)
  Hepatic function will be measured with a blood sample. Outcomes of interest include bilirubin, albumin, and total protein (all units: g/dL).
Difference in the incidence of Treatment-Emergent Adverse Events before and after supplementation as assessed by adverse events form | Pre-supplementation (12 wks), post-supplementation (12 wks)
  Adverse events will be recorded using the NIH's Adverse Events Form, ver 2.
Difference in the incidence of Treatment-Emergent Adverse Events before and after supplementation as assessed by checklist of changes to major organ systems | Pre-supplementation (12 wks), post-supplementation (12 wks)
  Common complaints of major organ system experienced over the last 3 days will be self-reported as present or not present for: stomachache, nausea, dizziness, coughing, wheezing, chest pain, weakness, increased headache, negative mood, rash, dry scalp, dry skin, nail changes, ear pain, decreased memory, itching, swelling, diarrhea, stiff joints, nose bleeds, heart burn, numbness, nasal congestion, ringing in ears, increased stress, decreased libido, constipation, shortness of breath, loss of appetite, loss of energy, blood in urine, & blood in stool.
Ability to comply with HMB supplementation as assessed by a daily diary & compliance check-ins | Post-supplementation (12 wks)
  Participants will complete a daily paper or electronic diary to document taking their supplement. Compliance checks will be conducted by the study staff via a call or email. Unused supplements will be counted at the end of the study. Compliance will be calculated as a percent (# of pills taken on time/total # of pills that should have been taken) x 100.
Ability to swallow HMB supplement as assessed by the PILL-5 survey | Week 1 of supplementation
  The PILL-5 survey is a 5 question survey that measures physical (e.g., pill sticks in my throat) and emotional (e.g., I have a fear of swallowing pills) swallowing ability. It will be self-reported using a 5-pt Likert scale (never, almost never, sometimes, almost always, always). A total score is calculated (range 0-20, with 20 representing maximum pill dysphasia).
Palatability of HMB supplement as assessed by the visual 5 faces hedonic scale | Week 1 of supplementation
  Whether participants like or dislike the taste of the supplement will be measured with a 5 faces hedonic scale with the numerical anchors ranging from 1 to 5 (best) and text anchors: dislike a lot; dislike a little; neither like nor dislike; like a little; like a lot.
Satisfaction of supplement dose volume as assessed by survey | Week 12 of supplementation
  A question will measure if participants felt the dose volume (number of tablets) were acceptable (yes or no).
Difference in satisfaction of supplement dose frequency as assessed by survey | Week 12 of supplementation
  A question will measure if participants felt the frequency (2 times per day) was acceptable (yes or no).

SECONDARY OUTCOMES:
Change in lower extremity strength with supplementation as assessed using a Biodex isokinetic system | Pre-supplementation (12 wks), post-supplementation (12 wks)
  Isokinetic dynamometry will be used to measure peak torque of hip extensors & flexors, knee extensors & flexors, and ankle plantarflexors and dorsiflexors (Newton-meters/body mass).
Change in muscle mass with supplementation as assessed by dual-energy x-ray absorptiometry (DXA) | Pre-supplementation (12 wks), post-supplementation (12 wks)
  Skeletal muscle mass (kg) will be measured using a whole body DXA scan.
Change in functional mobility with supplementation as assessed by the 10-meter walk test (10MWT) | Pre-supplementation (12 wks), post-supplementation (12 wks)
  The 10MWT will be performed at the participant's fastest walking speed over a 14-m walkway, with 2-m on each end for acceleration and deceleration. Time to travel the middle 10-m will be recorded by stopwatch and average speed (m/s) calculated. Usual orthoses and assistive devices will be permitted and used at each repeat assessment.
Change in functional mobility with supplementation as assessed by the Timed-up-and-go test (TUG) | Pre-supplementation (12 wks), post-supplementation (12 wks)
  The TUG will be performed at self-selected speed using a standard height chair with arms. Participants will stand up, walk 3-m, and return to their seat. Time (seconds) will be measured. Usual orthoses and assistive devices will be permitted and used at each repeat assessment.
Change in functional mobility with supplementation as assessed by the 6 minute walk test (6MWT) | Pre-supplementation (12 wks), post-supplementation (12 wks)
  The 6MWT will be performed at the participant's fastest walking speed on an indoor, oval walking path. Distance travelled (m) will be recorded and average speed (m/s) calculated. Usual orthoses and assistive devices will be permitted and used at each repeat assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States